CLINICAL TRIAL: NCT00002628
Title: PHASE I/II TRIAL OF THE ADDITION OF TAXOL TO THE HIGH DOSE CARBOPLATIN AND CYCLOPHOSPHAMIDE WITH AUTOLOGOUS PERIPHERAL BLOOD PROGENITOR CELL SUPPORT IN PATIENTS WITH BREAST CANCER
Brief Title: Addition of Paclitaxel to High-Dose Combination Chemotherapy in Treating Women With Metastatic Breast Cancer
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: St. Louis University (Other)
Organization: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: CDR0000064017; SLUMC-7915; NCI-V95-0608
Record Dates: First submitted 1999-11-01; First posted 2004-08-31 (Estimated); Last update posted 2014-01-10 (Estimated); Status verified 2000-04

CONDITIONS: Breast Cancer
Keywords: stage IV breast cancer; recurrent breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Filgrastim; Carboplatin; Cyclophosphamide; Mesna; Paclitaxel; Peripheral Blood Stem Cell Transplantation

INTERVENTIONS:
Biological: filgrastim
Drug: carboplatin
Drug: cyclophosphamide
Drug: mesna
Drug: paclitaxel
Procedure: peripheral blood stem cell transplantation

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining more than one drug may kill more tumor cells. Peripheral stem cell transplantation may be able to replace immune cells that were destroyed by chemotherapy used to kill tumor cells, allowing higher doses of chemotherapy to be used.

PURPOSE: Phase I/II trial to study the effectiveness of paclitaxel added to a regimen of high-dose chemotherapy with cyclophosphamide and carboplatin followed by peripheral stem cell transplantation in treating women with metastatic breast cancer.

DETAILED DESCRIPTION:
OBJECTIVES: I. Estimate the maximum tolerated dose of paclitaxel in combination with high-dose carboplatin/cyclophosphamide followed by autologous peripheral blood stem cell support in women with stage IV breast cancer. II. Assess the nonhematologic toxic effects associated with this combination. III. Assess the response rate, duration of response, and survival in chemotherapy-sensitive women with metastatic breast cancer treated with this regimen.

OUTLINE: This is a dose-finding study. All patients undergo collection of peripheral blood stem cells (PBSC) with granulocyte colony-stimulating factor (G-CSF) mobilization prior to high-dose chemotherapy. Cohorts of 3-5 patients are treated at successively higher dose levels of paclitaxel until a maximum tolerated dose (MTD) is found. Paclitaxel is given as a single 24-hour infusion, followed by fixed doses of high-dose cyclophosphamide for 2 days, then carboplatin for 4 days. Three days later, patients receive PBSC and G-CSF for hematopoietic reconstitution. Additional patients are entered at the MTD. Patients are followed every 3 months for 1 year, every 4 months for 1 year, and every 4-6 months thereafter.

PROJECTED ACCRUAL: 50 patients will be accrued. The study is expected to take 18 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically diagnosed, stage IV adenocarcinoma of the breast Previously untreated or prior adjuvant chemotherapy only CR or PR following 3-5 courses of induction chemotherapy for current diagnosis with one of the following: Cyclophosphamide/doxorubicin Cyclophosphamide/methotrexate/fluorouracil Cyclophosphamide/mitoxantrone No active CNS metastases on CT or MRI Hormone receptor status: Any status

PATIENT CHARACTERISTICS: Age: 18 to 65 Sex: Women Menopausal status: Pre- or postmenopausal Performance status: ECOG 0-2 Hematopoietic: WBC greater than 3,000 Platelets greater than 100,000 Hepatic: Bilirubin no greater than 2.0 mg/dL Renal: Creatinine clearance greater than 60 mL/min Cardiovascular: Left ventricular ejection fraction greater than 50% on MUGA or echocardiogram No abnormal cardiac conduction on EKG, i.e.: No second- or third-degree heart block No bundle-branch block No arrhythmia except: Supraventricular sinus tachycardia Occasional premature atrial or ventricular contractions Pulmonary: DLCO greater than 60% of predicted Other: No preexisting peripheral neuropathy No HIV antibody No history of second malignancy within 5 years except: Nonmelanomatous skin cancer Cervical carcinoma in situ No pregnant or nursing women

PRIOR CONCURRENT THERAPY: Biologic therapy: Not specified Chemotherapy: Hematologically recovered from prior chemotherapy Endocrine therapy: Failure on 1 prior hormonal regimen required for ER-positive disease (greater than 10 femtomoles) unless visceral metastatic crisis requires immediate chemotherapy Radiotherapy: Not specified Surgery: Not specified

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 1994-11

CONTACTS AND LOCATIONS:
Overall Officials: Paul J. Petruska, MD, Study Chair — St. Louis University
Locations (3):
- United States (3):
  - Indiana University Cancer Center, Indianapolis, Indiana
  - St. Louis University Health Sciences Center, St Louis, Missouri
  - Methodist Hospital-Central Unit, Memphis, Tennessee